CLINICAL TRIAL: NCT01039363
Title: Phase II Clinical Evaluation of Vorinostat Combined With Salvage Reinduction Chemotherapy Including Gemtuzumab Ozogamicin, Idarubicin and Cytarabine and Vorinostat Maintenance in Relapse or Refractory Acute Myeloid Leukemia Patients With 50 Years or Older
Brief Title: Vorinostat Combined With Gemtuzumab Ozogamicin, Idarubicin and Cytarabine in Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Dong Hwan (Dennis) Kim/Assistant professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-08-029
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2009-12-25 (Estimated); Status verified 2009-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: Relapse or refractory acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Idarubicin; Cytarabine; Vorinostat

ARMS (1):
- Vorinostat (Experimental): Vorinostat combined with salvage reinduction chemotherapy including Gemtuzumab ozogamicin, Idarubicin and Cytarabine and Vorinostat maintenance
  Interventions: Drug: Salvage reinduction chemotherapy including Gemtuzumab ozogamicin, Idarubicin and Cytarabine and Vorinostat

INTERVENTIONS:
Drug: Salvage reinduction chemotherapy including Gemtuzumab ozogamicin, Idarubicin and Cytarabine and Vorinostat — Salvage reinduction therapy:
  Vorinostat 200mg BID po (D1-14) Gemtuzumab ozogamicin 3 mg/m2 once (D1) Idarubicin 12mg/m2 for 2 days (D2-3) Cytarabine 500mg/m2 bid IV for 5 days (D2-6)
  Maintenance:
  Once achieved CR, then Vorinostat 200mg BID po for 2 weeks, then 1 week's rest (1 cycle) for 11 cycles
  * Vorinostat should be stopped at least 2 weeks ahead of starting of consolidation therapy.
  * Gemtuzumab will be omitted in a consolidation schedule.
  * Allogeneic hematopoietic stem cell transplantation (HSCT) can be performed if HLA-matched sibling or unrelated donor is available. Vorinostat will be stopped 2 weeks prior to starting of conditioning regimen for allogeneic HSCT.

SUMMARY:
The prognosis of elderly patients with relapsed or refractory acute myeloid leukemia (AML) is grave. Because of their chronological age and/or the presence of multiple co-morbidities, treatment-related mortality in elderly patients with AML is quite high although higher intensive treatment is mandatory to overcome chemoresistant characteristic of their disease. Several regimens have been evaluated as salvage chemotherapy for relapsed or refractory AML such as Mitoxantrone/High dose Cytarabine or Amsacrine/High dose Cytarabine. These regimens could achieve complete remission (CR) in a part of patients, but resulted in higher treatment related mortality (TRM). Accordingly, less intensive salvage regimen is needed for elderly patients with relapsed or refractory AML.

The activity of histone deacetylase (HDAC) inhibitor, Vorinostat or Suberoylanilide hydroxamic acid (SAHA), against AML has been suggested in cell line models and in animal model as well as in a phase 1 trial. The phase 1 study determined the MTD of oral Vorinostat as 200mg twice daily or 250mg thrice daily. In addition, the phase 1 trial showed the antitumor activity of Vorinostat with 17% of response rate in patients with advanced leukemia or myelodysplastic syndrome (MDS). Accordingly, further study is recommended to demonstrate the clinical activity of Vorinostat in AML.

In terms of the combining drug with Vorinostat, anthracycline is one of the best candidate. A in vitro study demonstrated that the combination of anthracycline (esp. idarubicin) with HDAC inhibitor have significant clinical activity against leukemia. Another candidate is Gemtuzumab ozogamicin, which is a calicheamicin-conjugated antibody directed against CD33 antigen on AML blasts. The U.S. FDA also approved the use of GO in relapsed AML as a monotherapy. A study also showed that the combinational therapy of GO with attenuated doses of standard induction chemotherapy could successfully induce CR without increasing treatment-related mortality in AML patients aged 55 or older. A in vitro study reported that HDAC inhibitor valproic acid augmented the clinical activity of GO toward CD33+ AML cells. The study demonstrated that the strategy using HDAC inhibitor together with GO could potentially induce synergistic proapoptotic activity against AML blasts without increasing toxicity. In our center, so far we treated relapsed or refractory AML patients using the salvage regimen including GO (3mg/m2/dayx1day) plus attenuated Idarubicin/Cytarabine (Idarubicin 12mg/m2/day for 2 days and intermediate dose Cytarabine). So far, the CR rate from the regimen is around 50% without increasing TRM. Accordingly, we will determine the efficacy and toxicity of Vorinostat-incorporating salvage regimen based on the GO+IA chemotherapy in patients 50 years old or older with relapsed or refractory AML.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 50 years.
2. ECOG Performance Status of 0, 1 or 2
3. Life expectancy of at least 12 weeks.
4. Subjects in relapse or refractory after any kinds of chemotherapy for acute myeloid leukemia expressing CD33 antigen on ≥ 50% of myeloblasts.
5. Adequate liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days and adequate bone marrow within 14 days prior to screening:

   1. Total bilirubin < 1.5 times the upper limit of normal
   2. ALT and AST < 2.5 x upper limit of normal
   3. Alkaline phosphatase < 4 x ULN
6. PT-INR/PTT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.]
7. Serum creatinine < 1.5 x upper limit of normal.
8. Signed and dated informed consent before the start of specific protocol procedures.

Exclusion Criteria:

1. History of cardiac disease: congestive heart failure >NYHA class 3 or 4; active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension.
2. History of HIV infection or chronic hepatitis B or C (except the case receiving Lamivudine or entecavir and in control of HBV infection)
3. Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
4. Patients with seizure disorder requiring medication (such as anti-epileptics)
5. Patients with evidence or history of bleeding diasthesis before diagnosis of acute myeloid leukemia
6. Patients undergoing renal dialysis
7. Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry.
8. Radiotherapy during study or within 3 weeks of start of study drug. (Palliative radiotherapy will be allowed). Major surgery within 4 weeks of start of study
9. Investigational drug therapy outside of this trial during or within 4 weeks of study entry
10. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
11. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study, such as Alzheimer's disease or dementia
12. Patients unable to swallow oral medications.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
response rate

CONTACTS AND LOCATIONS:
Overall Officials: Dong Hwan Kim, M.D.,Ph.D., Principal Investigator — Division of Hematology and Oncology/Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Garcia-Manero G, Yang H, Bueso-Ramos C, Ferrajoli A, Cortes J, Wierda WG, Faderl S, Koller C, Morris G, Rosner G, Loboda A, Fantin VR, Randolph SS, Hardwick JS, Reilly JF, Chen C, Ricker JL, Secrist JP, Richon VM, Frankel SR, Kantarjian HM. Phase 1 study of the histone deacetylase inhibitor vorinostat (suberoylanilide hydroxamic acid [SAHA]) in patients with advanced leukemias and myelodysplastic syndromes. Blood. 2008 Feb 1;111(3):1060-6. doi: 10.1182/blood-2007-06-098061. Epub 2007 Oct 25. PMID 17962510
- [Background] Bross PF, Beitz J, Chen G, Chen XH, Duffy E, Kieffer L, Roy S, Sridhara R, Rahman A, Williams G, Pazdur R. Approval summary: gemtuzumab ozogamicin in relapsed acute myeloid leukemia. Clin Cancer Res. 2001 Jun;7(6):1490-6. PMID 11410481
- [Background] Eom KS, Kim HJ, Min WS, Lee S, Min CK, Cho BS, Kim SY, Kim YJ, Lee DG, Choi SM, Cho SG, Kim DW, Lee JW, Shin WS, Kim CC. Gemtuzumab ozogamicin in combination with attenuated doses of standard induction chemotherapy can successfully induce complete remission without increasing toxicity in patients with acute myeloid leukemia aged 55 or older. Eur J Haematol. 2007 Nov;79(5):398-404. doi: 10.1111/j.1600-0609.2007.00946.x. Epub 2007 Oct 4. PMID 17916082
- [Background] Johnstone RW. Histone-deacetylase inhibitors: novel drugs for the treatment of cancer. Nat Rev Drug Discov. 2002 Apr;1(4):287-99. doi: 10.1038/nrd772. PMID 12120280
- [Background] Nimmanapalli R, Fuino L, Stobaugh C, Richon V, Bhalla K. Cotreatment with the histone deacetylase inhibitor suberoylanilide hydroxamic acid (SAHA) enhances imatinib-induced apoptosis of Bcr-Abl-positive human acute leukemia cells. Blood. 2003 Apr 15;101(8):3236-9. doi: 10.1182/blood-2002-08-2675. Epub 2002 Nov 21. PMID 12446442
- [Background] Sanchez-Gonzalez B, Yang H, Bueso-Ramos C, Hoshino K, Quintas-Cardama A, Richon VM, Garcia-Manero G. Antileukemia activity of the combination of an anthracycline with a histone deacetylase inhibitor. Blood. 2006 Aug 15;108(4):1174-82. doi: 10.1182/blood-2005-09-008086. Epub 2006 May 4. PMID 16675713
- [Background] ten Cate B, Samplonius DF, Bijma T, de Leij LF, Helfrich W, Bremer E. The histone deacetylase inhibitor valproic acid potently augments gemtuzumab ozogamicin-induced apoptosis in acute myeloid leukemic cells. Leukemia. 2007 Feb;21(2):248-52. doi: 10.1038/sj.leu.2404477. Epub 2006 Nov 23. PMID 17122863